CLINICAL TRIAL: NCT01371903
Title: The Effect of Patient Features on Opioid Induced End-Tidal CO2
Brief Title: The Effects of Patient Features on Opioid Induced End-Tidal CO2
Acronym: Capno
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Wayne Triner, Professor Emergency Medicine, Albany Medical College
Other Study IDs: 2792
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2011-06

CONDITIONS: Opioid Use During Medical Care
Keywords: morphine; fentanyl; dilaudid; opioid; capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Emergency department patients receiving opioid pain medicine such as morphine, fentanyl or Dilaudid are eligible. After medication exhaled carbon dioxide is measured. and recorded.

DETAILED DESCRIPTION:
Emergency department patients receiving opioid pain medicine such as morphine, fentanyl, or Dilaudid are eligible. After receiving the pain medication, a small soft plastic tube will be placed between the upper lip and nose. This tube is used to measure the amount of carbon dioxide the patient is breathing out. It can also be used to deliver oxygen if the provider feels the patient needs it. The carbon dioxide breathed out is measured and collected. Other information collected are height, weight, and vital signs. Patient participation time is approximately 2 hours during the emergency department visit.

ELIGIBILITY:
Inclusion Criteria:

* non intubated patients receiving intravenous opioid medications

Exclusion Criteria:

* mechanically ventilated patients
* patients with physiologic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving opioid such as morphine, fentanyl, or dilaudid during their emergency department visit.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
end tidal carbon dioxide | study start, 30 minutes, 60 minutes, 90 minutes, 120 minutes
  measured through small nasal cannula (plastic tube at base of nares)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Emergency Department, Albany, New York, United States